CLINICAL TRIAL: NCT06458777
Title: Evaluación de la Rentabilidad y Sensibilidad Del análisis automático Contra el análisis Manual de la poligrafía en el diagnóstico de Apnea Obstructiva Del sueño.
Brief Title: Evaluation of the Cost-Effectiveness and Sensitivity of Automatic Analysis Versus Manual Analysis of Polygraphy in the Diagnosis of Obstructive Sleep Apnea.
Status: Completed | Type: Observational
Sponsor: Hospital San Pedro de Logroño (Other)
Responsible Party: Sponsor
Other Study IDs: PI 608
Record Dates: First submitted 2023-08-02; First posted 2024-06-14 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with manual report of polygraphy
  Interventions: Diagnostic Test: poligraphy
- Patients diagnosed with automatical report of polygraphy
  Interventions: Diagnostic Test: poligraphy

INTERVENTIONS:
Diagnostic Test: poligraphy — OSA diagnosis

SUMMARY:
Obstructive sleep apnea (OSA) is a chronic pathology that affects more than 20% of the adult population. It is one of the main sleep disorders with great clinical, economic and social repercussions.

To assess the impact and severity of obstructive sleep apnea, the number of apneas and hypopneas per hour (AHI) is counted. To define that a person has OAS, a sleep study must have an AHI ≥15/h, predominantly obstructive, or the presence of an AHI ≥5/h accompanied by symptoms.

The diagnosis of certainty or exclusion, as well as the severity, is established with a sleep study. Polysomnography (PSG) continues to be the gold standard for the diagnosis of OSA, it encompasses the recording of cardiorespiratory and neurophysiological variables, which makes it possible to analyze sleep time and structure, the presence of different respiratory episodes and their repercussions. Respiratory polygraphy (RP) includes recording from a flow sensor, respiratory effort, oxygen saturation, heart rate, and also position but not EEG. There are several studies that have explored the diagnostic agreement of RP versus PSG, being a validated, useful and necessary test for the diagnosis of OSA in different clinical situations. Being cheaper and more accessible.

When talking about the diagnosis of OSA, it refers to establishing whether or not there is, the severity and the therapeutic decision that will greatly affect the quality of life, prognosis and day-to-day life of the patient, since it is a chronic disease.

It must be borne in mind that most studies are carried out in a field specialized in dream interpretation, so caution must be exercised in interpreting results in another field. PR teams incorporate increasingly better developed software that allows automatic analysis of records, but the technology and algorithms used vary depending on the device, and up to now the AASM continues to recommend manual analysis based on existing evidence. Several studies have examined the agreement between automatic and manual analysis of the PR record or between automatic analysis of PR and PSG. It seems that this agreement is reached above all in the highest AHIs, above 25-30, which may limit its use in clinical practice.

For this reason, it is important to carry out a study with a large number of patients to achieve statistical significance, and strong conclusions that support normal clinical practice, and to disable a study that does not meet the scientific requirements when interpreting and reading.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory polygraphs carried out at the San Pedro Hospital in the period of time between 2014-2020.
* Polygraphs corresponding to patients over 18 years of age.

Exclusion Criteria:

* Poor technical quality of polygraphy
* Patients with >50% central apnea or presence of Cheyne-Stokes respiration (CSResp).
* Lack of automatic and/or manual analysis of the polygraph.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dream Unit Patients with diagnostic suspicion of OSA
Sampling Method: Non-Probability Sample
Enrollment: 3144 (Actual)
Dates: Start 2014-01-19 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Cost-Effectiveness and Sensitivity of Automatic Analysis Versus Manual Analysis of Polygraphy in the Diagnosis of Obstructive Sleep Apnea. | 2 years
  effectiveness of the analysis described with the AHI (number of sleep apneas in each hour slept)
Evaluation of the Cost-Effectiveness and Sensitivity of Automatic Analysis Versus Manual Analysis of Polygraphy in the Diagnosis of Obstructive Sleep Apnea. | 2 years
  economic cost (measured in euros) of manual and automatic polygraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Pedro, Logroño, La Rioja, Spain

IPD SHARING:
Plan to Share IPD: Undecided